CLINICAL TRIAL: NCT02303886
Title: Evaluation of the Effects of Methylene Blue on Neuropathic Pain and Protein Biomarkers
Brief Title: Methylene Blue Intravenously and Chronic Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Adriana Miclescu, MD, PhD, DEAA, Uppsala University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NO8
Record Dates: First submitted 2014-11-16; First posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Methylene Blue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A Methylene blue 10 mg/ml 2mg/kg (Active Comparator): ten patients that recieved MB1 methylene blue 2 mg/kg infusion under 60 min
  Interventions: Drug: Methylene blue
- B Methylene blue 10 mg/ml 0.02 mg/kg (Placebo Comparator): Same patients received MB2 Methylene blue 0.02 mg/kg infusion under 60 min
  Interventions: Drug: Methylene blue

INTERVENTIONS:
Drug: Methylene blue — In NaCL0.9% 100 ml
  Other Names: methylthioninium chloride
Drug: Methylene blue — in NaCl 0.9% 100 ml
  Other Names: methylthioninium chloride

SUMMARY:
Aim of Investigation Methylene blue (MB) is a diaminophenothiazine with antioxidant, anti-inflammatory properties and with inhibitory effects on nitric oxide. The aim of this study was to determine the clinical effectiveness of MB in the treatment of neuropathic pain.

Methods Ten patients with neuropathic pain were randomized to receive one of the two treatments: methylene blue (MB1) 2 mg/kg (10 mg/mL Methyltioninklorid, Apoteket, Umeå, Sweden) or methylene blue (MB2) 0.02 mg/kg. Both MB solutions were infused intravenously over 60 minutes. The sensory function and the pain were evaluated at baseline and at 60 min after the start of infusions. A pain journal was kept by the patients in the following 5 days. Plasma and urinary concentrations of 8-isoprostane-prostaglandin F2α (8-iso-PGF2α) an indicator of oxidative injury, were measured with radioimmunoassay (RIA). A panel of 92 proteins biomarkers were determined with Proximity Extension Assay (PEA) prior and after infusions.

comparison with the control group. MB infusion produced an enhancement of prolactin.

DETAILED DESCRIPTION:
Patients Study participants were screened from a pool of patients with chronic treatment resistant neuropathic pain and were eligible to participate in the study after giving written informed consent Study design The patients visited the Pain Clinic twice. Oral and written information about the study was provided and informed consent obtained. Demographic data (date of birth, sex, and ethnic background, medical and surgical history) were recorded. Information about the patients' assessments were recorded before the injection, including current medication and other (successful or non-successful) treatment attempts. The same investigator (AM) performed all study procedure assessments. Assessments of sensory function were performed before drug administration.

Administration of study drug Ten patients were randomized by a computer generated random list to receive either methylene blue 2mg/kg (10 mg/mL Methyltioninklorid, Apoteket, Umeå, Sweden) or methylene blue 0.02 mg/kg (that served as control), both infused intravenously over 60 minutes. After monitors for electrocardiography, noninvasive arterial blood pressure, and pulse oximetry were attached, a dedicated 20-gauge cannula was inserted into the dorsum of the nondominant hand for administration of the study drugs. The pain was measured at baseline and at 60 min after the start of infusion (NRS scale) and also with a pain diary during the next 24 hours and the following 5 days. ECG, pulse, blood pressure, O2 saturation, were continuously recorded during the infusion. Blood and urine samples were taken before and after the infusion of MB. Neither the subjects of the experiment nor the person examining the patients knew the concentration of MB in the infusion. The infusions of methylene blue in sterile saline (NaCl 0.9%) were prepared by another person who had access to the randomization list but not involved in the monitoring of the patients. The infusions bags were covered in opaque red wrappes and the infusions sets were opaque.

Pain Assessment were performed Before and after MB administration, Evaluation of sensory function was performed using bedside examination according to EFNS guidelines: light touch, pinprick sense, warmth (40°) and cold (25°) temperature stimuli were tested. The contralateral uninjured side served as within-patient control. The patient compared the sensations in both between sides and reported if there was any hypoesthesia, hyperesthesia, allodynia or simply normal sensations to the different stimuli. The pain recordings were determined before and after infusion of MB. Patients kept a diary where they could pick their pain levels on a scale between 0 and 10 (NRS) at every 6 hours after the infusion in the first 24 hours and at 8 hours in the next 5 days.

Peripheral venous blood was drawn from fasting subjects using a 19-gauge needle. Urine was collected into additive-free tubes. Plasma was prepared from blood collected into tubes containing heparin by centrifugation (3500x g for 12 min). Urine and plasma samples were stored at -70◦C until analysis. Blood and urine samples were collected before and after the infusion of MB.

Plasma and urine concentrations of isoprostane 8-iso-PGF2 alpha (an indicator of oxidative injury),Proximity Extension Assay (PEA) has been found to have specificity of detection and analysis of an increased range of target molecules. PEA technology involved in this study a panel of 92 oligonucleotide labeled antibody probe pairs (Proseek assay kit), Non-parametric statistical methods were performed by the author with GraphPad PRISM 5.0 (GraphPad Software, La Jolla, San Diego, CA, www.graphpad.com 5.0). Data are presented as mean and SD with 95% confidence intervals. The level of significance was set at a p value <.05.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects > 18 years of age
* Be able to understand and comply with the requirements of the study
* Patients with a history of persistent peripheral and central neuropathic pain interfering with daily activities of at least 3 months duration
* Patients with previous unsuccessful treatment of neuropathic pain
* Spontaneous or evoked pain upon standardized test (mechanical, movement)> 50 on a 100 mm VAS scale
* Informed written consent

Exclusion Criteria:

* Any condition that may confound assessment of pain (acute pain)
* Any condition/disease that could interfere with the study measurements, e.g. peripheral vascular disease, diabetes mellitus, alcohol/opioids addiction
* Noncooperation, insufficient Swedish language
* Treatment with antidepressants, antiepileptics, opioids, lidocaine patches was not accepted the day before and the day of the visit
* Pregnancy
* Treatment with NO releasing drugs, anti-cytokine therapy
* Diabetes mellitus type I, malignancy, increased pulmonary hypertension, cardiac ischemic disease, decreased glomerular filtration rate<30 ml/min, decreased liver function, Glu-6-PDH deficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Pain (visual analogue scale) | 60 min, every 6 hours after the infusion in the first 24 hours and at 8 hours in the next 5 days
  VAS

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Miclescu, Principal Investigator — Uppsala University Hospital